CLINICAL TRIAL: NCT00452491
Title: A Cohort of Pre-pubertal Children for the Study of Optimization of Methods of Administration of the Biosynthetic Growth Hormone MAXOMAT ® in the Treatment of Severe Early Onset Intrauterine Growth Retardation
Brief Title: MAXOMAT ® in the Treatment of Severe Early Onset Intrauterine Growth Retardation on Pre-pubertal Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH5126A
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: somatropin
- 2 (Active Comparator)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 0.2 IU/kg/day 7 days per week given sequentially (alternating periods of 6 months of treatment and 6 months of no treatment) for 3 years
  Arms: 1
Drug: somatropin — 0.2 IU/kg/day 7 days per week given continuously for 3 years
  Arms: 2

SUMMARY:
1. To test for equivalence in terms of catch-up growth between the 2 therapeutic regimens
2. To specify the best period of treatment
3. To assess the efficacy of treatment based on final adult height of these children

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubertal children of either sex presenting with severe early onset intrauterine growth retardation (I.U.G.R.)
* Height Less Than or Equal to -3 SD

Exclusion Criteria:

* Age less than 3 years

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 1993-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Efficacy data : measurement of height | at trimestrial visit

SECONDARY OUTCOMES:
laboratory test assessment and evaluation of bone age | at every other visit
measurement of anti-GH and anti-ECP antibodies | one visit out of four
Tolerance data : undesirable events | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Marie SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France